CLINICAL TRIAL: NCT04775589
Title: Telehealth Stepped Exercise Program for Rural Veterans With Knee Osteoarthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15997
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis
Keywords: Exercise; Physical Therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stepped Exercise for Knee Osteoarthritis (Experimental): Patients start with a home-based exercise program, supported by an internet-based tool (Step 1). Patients are then assessed for degree of improvement in symptoms, and then can step up sequentially to telephone or video-based physical activity coaching (Step 2) and physical therapy (Step 3) if they do not make clinically relevant improvements in prior steps.
  Interventions: Behavioral: Stepped Exercise for Knee Osteoarthritis

INTERVENTIONS:
Behavioral: Stepped Exercise for Knee Osteoarthritis — Patients start with a home-based exercise program, supported by an internet-based tool (Step 1). Patients are then assessed for degree of improvement in symptoms, and then can step up sequentially to telephone or video-based physical activity coaching (Step 2) and physical therapy (Step 3) if they do not make clinically relevant improvements in prior steps

SUMMARY:
The goal of this study is to evaluate a telehealth Stepped Exercise Program for Knee OsteoArthritis (STEP-KOA) among rural veterans. Methods: This is a single arm, pre-post pilot trial of the 6-month STEP-KOA program among rural Veterans with a physician diagnosis of knee OA who self-report knee pain ≥3 on a 0-10 scale and self-reported difficulty with either walking or stair climbing. We aim to enroll 20 Veterans in this project but may enroll up to 30 in order to obtain sufficient information to evaluate the program, particularly among Veterans who live in very rural areas. Assessments will be conducted via a combination of telephone and video at baseline and 2-, 4-, and 6-month follow-up. Assessments will include questionnaires related to pain, function and physical activity, as well as several physical performance tests. STEP-KOA begins with a low cost, primarily self-directed exercise program (supported by an internet-based tool; Step 1). Patients are then assessed for degree of improvement in symptoms, and then can step up sequentially to telephone or video-based physical activity coaching (Step 2) and physical therapy (Step 3) if they do not make clinically relevant improvements in prior steps. For this project, patients will be assessed approximately every 2 months to determine step progression. Participants will advance to the next step if they do not meet response criteria for pain and function established by the Outcome Measures in Rheumatology group and the Osteoarthritis Research Society International (OMERACT-OARSI). The Step 2 intervention involves bi-weekly telephone or video calls. Step 3 involves 3 telehealth PT visits, based on standard care for knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Rural dwelling Veterans (VA healthcare users)
* Clinician diagnosis of knee osteoarthritis
* Self-reported knee pain =>3 on a scale of 0-10 and self-reported difficulty either walking or stair climbing.

Exclusion Criteria:

* Advanced Dementia
* Psychosis
* Active substance abuse disorder
* Meniscus or ACL tear in the past 6 months
* Total joint replacement or other major lower extremity surgery in the past 6 months
* Severe hearing or visual impairment (e.g. unable to participate in STEP-KOA intervention components)
* Serious / terminal illness
* Unstable angina
* History of ventricular tachycardia
* Unstable chronic obstructive pulmonary disease (two hospitalizations within the previous 12 months and/or on oxygen)
* Uncontrolled hypertension (diastolic blood pressure >110 mm/Hg or systolic > 200mm/Hg)
* Stroke with moderate to severe aphasia
* Recent history of falls
* Resident of a long-term care facility
* Hospitalization for a cardiovascular condition in the past 3 months
* Other health conditions that would make home exercise unsafe or participation in the program not feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index | Baseline to 6 months
  24-item measure assessing lower extremity pain, stiffness and function. All items are measured on a 5-point Likert scale (0-4; total score 0-96), with higher scores indicating worse symptoms.

SECONDARY OUTCOMES:
30-second chair stand test | Baseline to 6 months
  Participants are asked to rise and sit back down in a chair as many times as they can during 30 seconds, without using hands or arms for support. Higher numbers of chair stands indicate better function.
2 minute march test | Baseline to 6 months
  Participants are asked to march in place, taking as many "steps" as they can within 2 minutes, bringing the knees to approximately a 90-degree angle. If the patient is not bringing knees to an appropriate height, the study team member administering the test will ask them to raise their knees higher; if proper knee height cannot be maintained, the patient may continue the test, but this is noted on the score sheet. Higher numbers of steps indicate better function.

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Allen, PhD, Principal Investigator — Durham VAMC
Locations (1):
- Durham VA Healthcare System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No